CLINICAL TRIAL: NCT04155801
Title: An Open-Label, Multicenter Study to Assess the Efficacy and Safety of Salix Probiotic Blend in Subjects With Functional Gastrointestinal Disturbances
Brief Title: A Study to Assess the Efficacy and Safety of Salix Probiotic Blend in Participants With Functional Gastrointestinal Disturbances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PBGD1001
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Functional Gastrointestinal Disorders
Keywords: Gastrointestinal Disorders, Functional
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Salix Probiotic Blend (Experimental): Participants will receive a Salix Probiotic Blend capsule orally once a day for 30 days.
  Interventions: Dietary Supplement: Salix Probiotic Blend

INTERVENTIONS:
Dietary Supplement: Salix Probiotic Blend — Oral capsule. The probiotic strains comprise the Salix Probiotic Blend include 3 strains of Bifidobacterium lactis (Bl-04®, Bi-07®, HN019) and 2 strains of lactobacillus (Lactobacillus acidophilus [NCFM]® and Lactobacillus paracasei [Lpc-37]®).

SUMMARY:
The primary objective of this study is to assess the safety and efficacy of Salix Probiotic Blend, administered orally for 30 days, in participants with functional gastrointestinal (GI) disturbances.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have symptoms of GI disturbances.
* Participant has recurrent abdominal pain, discomfort, bloating, and/or abdominal distention associated with a change in the frequency of stool and/or a change in the form (appearance) of stool.
* Participant is able to understand the nature and purpose of the study and provide informed consent.
* Sexually active males and sexually active females of child-bearing potential, defined as neither surgically sterile nor post-menopausal (that is, females age >45 years and no menstrual periods for at least 1 year), must agree to use a highly effective method of contraception from Screening to 30 days post last dose of study product. Acceptable forms of contraception include the following:

  * Abstinence
  * Oral, injected, or implanted hormonal methods of contraception
  * Intrauterine device or intrauterine contraceptive system
  * Condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository
  * Female whose last sexual intercourse with males was ≥6 months post-vasectomy

Exclusion Criteria:

* Participant has active or a history of inflammatory bowel disease.
* Participant has other significant systemic diseases such as active cancer therapy, active/ongoing infection, uncontrolled diabetes, chronic renal failure, cirrhosis, congestive heart failure, and severe Chronic Obstructive Pulmonary Disease (COPD).
* Participant has used antipsychotic medications within 3 months prior to Screening.
* Participant has used systemic steroids within the month prior to Screening.
* Participant has suffered from a major psychiatric disorder within the past 2 years.
* Participant is pregnant or breastfeeding.
* Participant has a known lactose intolerance.
* Participant is immunocompromised or has an immunodeficiency syndrome of any kind.
* Participant has undergone any abdominal surgery, except for hernia repair or appendectomy.
* Participant has had active treatment with prescription medication for irritable bowel syndrome (IBS) within 6 weeks prior to Screening.
* Participant has been diagnosed with infectious gastroenteritis within 1 month prior to Screening.
* Participant has undergone treatment with probiotics within 6 weeks prior to Screening.
* Participant is on active treatment with antibiotics.
* Participant has a known fructose intolerance.
* Participant is currently on a low fermentable oligo-, di-, mono-saccharides and polyols (FODMAP) diet.
* Participant has a known diagnosis of gastroparesis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with a Positive Response to the Product Satisfaction Question | Day 42 (End of Study [EOS] Visit)
  Participants will be asked to consider how they felt in the past week in regard to their gastrointestinal well-being and symptoms of abdominal discomfort or pain, bloating, or distension, gas, and altered bowel habit, and to respond to the following overall product satisfaction question: "Compared to the way you felt before beginning the supplement, how strongly do you feel you have had improvement of your overall gastrointestinal well-being?". Responses will be assessed on a Likert 6-point scale. Potential responses will include 1=strongly agree, 2=disagree, 3=slightly disagree, 4=slightly agree, 5=agree, and 6=strongly agree. The percentage of participants with the response of 4=slightly agree, 5=agree, and 6=strongly agree will be reported.

SECONDARY OUTCOMES:
Measures of Quality of Life Using the Irritable Bowel Syndrome Quality of Life (IBS-QOL) Questionnaire | Baseline up to Day 42 (EOS Visit)
  To assess quality of life prior to and post-treatment, participants will be asked to rate 34 quality of life questions from the sub-categories of dysphoria, interference with activity, body image, health worry, food avoidance, social reaction, sexual, and relationship, using the following scale: 1=Not at all; 2=Slightly, 3=Moderately; 4=Quite a bit; 5=Extremely. Lower scores=better IBS-related QoL.
Severity of Diarrhea, Constipation, Straining, Urgency, Abdominal Pain/Discomfort, Bloating, and Distention as Measured by the Gastrointestinal (GI) Health Symptom Questionnaire | Baseline up to Day 42 (EOS Visit)
  Participants will be asked to rate GI symptoms of diarrhea, constipation, straining (difficulty) to move bowels, urgency to move bowels (need to rush to the bathroom to avoid an accident), abdominal pain/discomfort, bloating, and distention (abdominal swelling), using a severity scale where 0 represents "none" and 10 represents "severe".
Frequency of GI Symptoms as Measured by the GI Health Symptom Questionnaire | Baseline up to Day 42 (EOS Visit)
  Participants will be asked to report the number of days per week (that is, never, 1-2 days, 3-4 days, 5-6 days, or 7 days) they experienced the symptoms of diarrhea, constipation, straining (difficulty) to move their bowels, urgency to move their bowels (need to rush to the bathroom to avoid an accident), abdominal pain/discomfort, bloating, distention (abdominal swelling), ability to fully empty bowels, and excessive passage of gas.
Satisfaction with Ability to Fully Empty Bowels as Measured by the GI Health Symptom Questionnaire | Baseline up to Day 42 (EOS Visit)
  Participants will be asked to rate how satisfied they are with the ability to fully empty their bowels on a scale where 0 represents "not satisfied" and 10 represents "very satisfied".
Passage of Gas Symptoms as Measured by the GI Health Symptom Questionnaire | Baseline up to Day 42 (EOS Visit)
  Participants will be asked to rate their excessive passage of gas symptoms on the scale where 0 represents "never" and 10 represents "frequently".
Satisfaction with Bowel Habits as Measured by the GI Health Symptom Questionnaire | Baseline up to Day 42 (EOS Visit)
  Participants will be asked to rate how satisfied they are with their bowel habits on a scale where 0 represents "not satisfied" and 10 represents "very satisfied".
Overall Product Satisfaction Evaluation | Day 30
  Participants will be asked to respond to the statement "Taking everything into consideration, would you say you are satisfied with this probiotic supplement, overall?" with a response of "Yes", "No", or "Do Not Know".
Change From Baseline in Intestinal Fatty-Acid Binding Protein (I-FABP) Levels (Intestinal Integrity Serum Marker) at Day 30 | Day 30
  Intestinal permeability assessments will be conducted through the evaluation of serum I-FABP levels in a blood sample collected from participants at Baseline and Day 30.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Mathew, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Bausch Site 001, San Antonio, Texas, United States